CLINICAL TRIAL: NCT06682013
Title: A Randomized Pilot Study Comparing the Feasibility of Using a Virtual Agent vs. an Off-site Human Agent to Onboard Oncology Patients to a Remote Monitoring Device
Brief Title: Virtual Agent Feasibility in Oncology Patients (NTT Data)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00116186
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — reducing agent and tunicamycin-responsive protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virtual agent (Experimental)
  Interventions: Device: Virtual agent
- Human agent (Active Comparator)
  Interventions: Other: Human agent

INTERVENTIONS:
Device: Virtual agent — The virtual agent is an interactive audio agent that is similar to voice agents that interact with callers in many industries today. They create a very human-like interaction in contrast to more traditional virtual call agents that can only respond to menu options (e.g. "choose "1" for appointments, choose "2" for questions about your bill", etc.). The virtual agent is engineered to accomplish the very specific task of onboarding the patient on use of the RPM devices. It is trained to understand normal human English speech, detects emotional tone and frustration of callers, and is trained to deescalate when appropriate.
  Arms: Virtual agent
Other: Human agent — The human agent will onboard the patient on use of the RPM devices.
  Arms: Human agent

SUMMARY:
The purpose of this study is to compare the use of a virtual agent vs. a human agent when onboarding oncology patients over the telephone to Remote Patient Monitoring (RPM) devices. RPM devices are instruments that a patient can use to measure their own weight and vital signs. Both the virtual and human agents will be available by telephone to instruct the patient on how to use the RPM devices to measure weight, blood pressure, heart rate, temperature, and oxygen saturation. Patients will be randomized to either the virtual or human agent, have assessments of their medical and oncological history, overall well-being, body measurements, and vital signs, and will complete questionnaires about their experience.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.
2. Age ≥18
3. Cancer (solid tumor)
4. Planning to return to Duke Cancer Center clinic for three days in a row

   * Patients whose treatment does not require that they return to clinic for three days in a row, but who are willing to voluntarily return to participate in this study are permitted to enroll.
5. Eastern Cooperative Oncology Group (ECOG) score of 0-2
6. Native fluency of spoken English as determined by the investigator

   * Non-native English speakers are permitted to enroll if they have achieved native fluency.
7. Vitals as collected by the clinic using Duke maintained equipment must be within the ranges specified by the remote patient monitoring devices.

   * Weight ≤ 180 kg
   * Systolic blood pressure ≤ 300 mmHg
   * Pulse rate of 40-200 bpm
   * SpO2 of 70-100%
   * Temperature 34.0-42.2°C
8. Arm circumference of 22-42 cm

Exclusion Criteria:

1. 1. Vision, speech, auditory, physical, cognitive or other impairment that has the potential to interfere with the use of the remote patient monitoring device or agent, in the opinion of the investigator or study coordinator.
2. Has an implanted pacemaker, arterio-venus (A-V) shunt, a history of mastectomy or lymph node clearance, history of severe blood flow problems or blood disorders, or a history of severe circulatory deficit in the arm.
3. Is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Usability of virtual agent vs. human agent for onboarding patients to RPM devices as assessed by the System Usability Scale (SUS) | Day 1, Day 2, Day 3
  The SUS is a questionnaire that assesses perceived usability. It includes 10 five-point items with alternating positive and negative tone. The final score is a number 0-100 with a higher score indicating better usability.

SECONDARY OUTCOMES:
Description of the patient experience when using a virtual agent in the context of teaching a patient as assessed by the patient experience survey. | Day 3
  The patient experience survey includes 3 open-ended questions about experience with the training process, input on using monitoring devices at home, and any other important information for the researchers to know. Descriptive analysis will be conducted within each arm.
Identification of opportunities to improve the use of a virtual agent in the context of teaching a patient as assessed by the patient experience survey. | Day 3
  The patient experience survey includes 3 open-ended questions about experience with the training process, input on using monitoring devices at home, and any other important information for the researchers to know. Descriptive analysis will be conducted within each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Alder, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No